CLINICAL TRIAL: NCT06562127
Title: TBI Rehabilitation and Activation in Veterans (TRAIN-Vets)
Brief Title: TBI Rehabilitation and Activation in Veterans
Acronym: TRAIN-Vets
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Northern California Institute of Research and Education (Other)
Collaborators: San Francisco Veterans Affairs Medical Center (U.S. Federal Agency); VA Palo Alto Health Care System (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HT9425-24-1-0720; HT9425-24-1-0720 (Other Grant/Funding Number: Department of Defense)
Record Dates: First submitted 2024-07-18; First posted 2024-08-20 (Actual); Last update posted 2025-05-16 (Actual); Status verified 2025-05

CONDITIONS: Traumatic Brain Injury
Keywords: Cognition; Cognitive training; Physical exercise; Head injury; Traumatic brain injury
MeSH Terms: conditions — Brain Injuries, Traumatic; Motor Activity; Craniocerebral Trauma

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- TRAIN-Vets (Experimental): TRAIN-Vets is an 8-month intervention with aquatic-based exercise training and cognitive training combined with personalized dementia risk factor reduction sessions. This intervention entails 6 months of thrice-weekly aquatic-based exercise training at Veterans Affairs Palo Alto Health Care System (VAPAHCS). After completion of the 6-months of exercise training, Veterans in this condition will participate in 2 months of weekly structured on-line cognitive training focused on improvement of executive function and attention based out of the San Francisco Veterans Affairs Health Care System (SFVAHCS). Concurrently, Veterans in TRAIN-Vets will also participate virtually in personalized risk factor reduction sessions based at SFVAHCS focused on other risk factors and symptoms.
  Interventions: Behavioral: TRAIN-Vets
- Health Education Control (Other): The Health Education Control (HEC) receives mailed educational materials about brain health and dementia risk factor reduction over 8 months, as well as regular contact with study staff.
  Interventions: Behavioral: Health Education Control

INTERVENTIONS:
Behavioral: TRAIN-Vets — The TRAIN-Vets intervention entails 6 months of thrice-weekly aquatic-based exercise training at Veterans Affairs Palo Alto Health Care System (VAPAHCS). After completion of the 6-months of exercise training, Veterans in this condition will participate in 2 months of weekly structured on-line cognitive training focused on improvement of executive function and attention based out of the San Francisco Veterans Affairs Health Care System (SFVAHCS). Concurrently, Veterans in TRAIN-Vets will also participate virtually in personalized risk factor reduction sessions based at SFVAHCS focused on other risk factors and symptoms.
  Arms: TRAIN-Vets
Behavioral: Health Education Control — The Health Education Control (HEC) receives mailed educational materials about brain health and dementia risk factor reduction over 8 months, as well as regular contact with study staff.
  Arms: Health Education Control

SUMMARY:
This trial will evaluate the impact of a multicomponent program (TBI Rehabilitation and Activation in Veterans; TRAIN-Vets) on improving cognitive function over an 8-month trial period in older Veterans with traumatic brain injury (TBI). Older Veterans with a history of TBI and subjective cognitive complaints will be enrolled and randomly assign to either the TRAIN-Vets intervention (consisting of aquatic-based exercise training, cognitive training, and lifestyle coaching) or the Health Education Control, where they will receive educational materials about brain health and healthy lifestyles.

DETAILED DESCRIPTION:
The purpose of the proposed trial is to evaluate the impact of a multicomponent training program (TRAIN-Vets) on improving cognitive function and other outcomes over an 8-month period in older Veterans with TBI and cognitive complaints. The primary aim of the trial is to evaluate the efficacy of the TRAIN-Vets intervention to improve cognitive function in Veterans with TBI. Secondary aims of the proposed research are to evaluate the efficacy of TRAIN-Vets to improve: 1) individual cognitive domain scores, 2) psychological and social measures (sleep, mood, social and community engagement, diet, and life satisfaction), and 3) physical fitness.

The investigators will randomize 120 older Veterans with TBI and cognitive complaints aged 50 or older to TRAIN-Vets or Health Education Control (HEC). Participants randomized to the TRAIN-Vets group will engage in aquatic-based exercise training and cognitive training combined with personalized risk factor reduction related to their brain health risk factors. This intervention entails 6 months of thrice-weekly aquatic-based exercise training at Veterans Affairs Palo Alto Health Care System (VAPAHCS). After completion of the 6-months of exercise training, Veterans in this condition will participate in 2 months of weekly structured on-line cognitive training focused on improvement of executive function and attention based out of the San Francisco Veterans Affairs Health Care System (SFVAHCS). Over the 8 months, Veterans in TRAIN-Vets will also participate virtually in monthly personalized risk reduction sessions based at SFVHCS focused on improving other risk factors and symptoms. Participants in the HEC group will be mailed educational materials about brain health and dementia risk factor reduction throughout the 8 months. HEC participants will be contacted monthly through phone calls to check in and maintain interest. All participants will complete a phone screening, baseline in person and virtual visits, and follow-up visits with blinded assessors (to assess outcomes) at approximately 6 and 8 months.

ELIGIBILITY:
Inclusion Criteria:

* Veteran, age 50-89 years
* History (more than 6 months post injury) of mild or moderate TBI defined by the Ohio State University TBI Identification Method and DOD/VA Clinical Practice Guidelines for Definition of TBI
* Sufficient vision and hearing to allow cognitive testing
* Willingness to participate in water-based exercise program + cognitive training program for eight months
* Approval of primary medical provider to participate in a water-based exercise program
* Subjective cognitive complaints as evidenced by self-report
* English proficiency to allow for cognitive testing
* Internet connected device to participate in testing and cognitive training

Exclusion Criteria:

* Current severe and unstable psychiatric disorder
* Diagnosis of dementia, Montreal Cognitive Assessment score less than 18, or delirium
* TBI within the past 6 months
* Acute illness or unstable chronic illness
* Current severe cardiac disease
* Severe TBI or open head injury
* Inability to exercise consistently
* Inability to read, verbalize understanding, and voluntarily sign the Informed Consent

Ages: 50 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2025-05-12 (Actual); Primary Completion 2028-02 (Estimated); Study Completion 2028-02 (Estimated)

PRIMARY OUTCOMES:
Cognitive Change (Composite Score) | 8 months
  Change in global composite score calculated from the z-scores from all cognitive measures [Wechsler Adult Intelligence Scale, 4th edition (WAIS-IV) Digit Span Forward, WAIS-IV Digit Span Backwards, WAIS-IV Digit Span Sequencing, Trail Making Test A and B; Delis-Kaplan Executive Function System (DKEFS) Stroop Inhibition Time & Errors; DKEFS Stroop Inhibition-Switching Time & Errors; DKEFS Verbal Fluency Switching; Benson Figure Copy and Recall; Hopkins Verbal Learning Test (HVLT) Learning and Delayed Recall Trials]. The total score is reported. Higher values signify higher cognitive performance. A z-score of 0 represents the population mean.

SECONDARY OUTCOMES:
Cognitive Sub-Domain Change: Executive Function (Composite Score) | 8 months
  Change in executive function composite score calculated from the z-scores from all executive function measures (WAIS-IV Digit Span Sequencing, DKEFS Color-Word Interference (Stroop) Inhibition, Trails B, DKEFS Verbal Fluency Switching, DKEFS Stroop Inhibition-Switching). The total score is reported. Higher values signify higher executive function performance. A z-score of 0 represents the population mean.
Cognitive Sub-Domain Change: Learning/Memory (Composite Score) | 8 months
  Change in learning/memory composite score calculated from the z-scores from all learning/memory measures (HVLT learning and delayed recall and Benson Figure recall). The total score is reported. Higher values signify higher learning/memory performance. A z-score of 0 represents the population mean.
Targeted Risk Factor Change (Composite Score) | 8 months
  Change in targeted risk factor composite score calculated from the z-score from all risk factor measures [sleep quality (Pittsburgh Sleep Quality Inventory), mood (Patient Health Questionnaire - 9), social and community engagement (PROMIS Satisfaction with Participation in Discretionary Social Activities), and diet (MIND Diet Questionnaire)]. The total score is reported. Higher values signify more favorable risk factors. A z-score of 0 represents the population mean.
Quality of Life Change | 8 months
  Change in life satisfaction (Satisfaction with Life Scale). Higher score indicates better quality of life; range = 5 to 35.
Physical Fitness Change | 8 months
  Change in peak VO2, or VO2Max, defined as the minute volume of O2 utilization.

CONTACTS AND LOCATIONS:
Overall Officials: Kristine Yaffe, MD, Principal Investigator — University of California, San Francisco
Locations (2):
- United States (2):
  - VA Palo Alto Health Care System, Palo Alto, California
  - San Francisco VA Health Care System, San Francisco, California

IPD SHARING:
Plan to Share IPD: No